CLINICAL TRIAL: NCT06394986
Title: Cardio-fistular Recirculation in Patients With Chronic Heart Failure and Preserved Left Ventricle Ejection Fraction
Status: Completed | Type: Observational
Sponsor: Moscow Regional Research and Clinical Institute (MONIKI) (Other Government)
Responsible Party: Principal Investigator, Alexey Zulkarnaev, Leading Researcher in Surgical Department of Kidney Transplantation, Moscow Regional Research and Clinical Institute (MONIKI)
Other Study IDs: ABZ_310518
Record Dates: First submitted 2024-04-29; First posted 2024-05-01 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Chronic Kidney Disease 5D; Heart Failure; Heart Failure NYHA Class I; Heart Failure NYHA Class II
Keywords: arteriovenous fistula; hemodialysis; cardiac output; heart failure; volume blood flow; cardio-fistular recirculation; cardiopulmonary recirculation; ejection fraction
MeSH Terms: conditions — Heart Failure; Arteriovenous Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group
  Interventions: Procedure: Hemodialysis session

INTERVENTIONS:
Procedure: Hemodialysis session — Change of arteriovenous fistula volume blood flow / cardiac output ratio in patients with chronic heart failure (NYHA I-II classes) and with preserved ejection fraction as a result of a hemodialysis session will be explored.

SUMMARY:
This is a single-arm cohort study aimed to evaluate change of arteriovenous fistula volume blood flow / cardiac output ratio in patients with chronic heart failure (NYHA I-II classes) and with preserved ejection fraction as a result of a hemodialysis session after a "long" interdialysis interval.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent,
* > 18 years
* maintenance ("chronic") hemodialysis,
* native arteriovenous fistula,
* arteriovenous fistula volume blood flow ≥1 l/min,
* arteriovenous fistula volume blood flow / cardiac output ratio < 0.3,
* interdialysis weight gain <5% of "dry" body weight,
* sufficient hemodialysis dose (eKt/V > 1.2),
* chronic heart failure (NYHA I-II classes only),
* preserved left ventricular ejection fraction (≥50%),
* absence of arrhythmias (except first-degree atrioventricular block block),
* absence of heart valve disease (except mitral regurgitation grade I-II),
* absence of intradialysis hypo/hypertension
* "long" interdialysis interval (3 days).

Exclusion Criteria:

* hypo/hypertension during or after hemodialysis,
* arrhythmias (except first-degree atrioventricular block) after hemodialysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stable adult patients on maintenance hemodialysis.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2019-02-18 (Actual); Study Completion 2019-02-18 (Actual)

PRIMARY OUTCOMES:
Change in cardio-fistular recirculation | One hour before and two hours after the hemodialysis session.
  Change in arteriovenous fistula volume blood flow / cardiac output ratio

CONTACTS AND LOCATIONS:
Overall Officials: Alexey B Zulkarnaev, MD, Prof., Principal Investigator — Moscow Regional Research and Clinical Institute (MONIKI)
Locations (1):
- Moscow Regional Research and Clinical Institute (MONIKI), Moscow, Russia